CLINICAL TRIAL: NCT02519283
Title: Get With the Guidelines in ED Patients With Heart Failure
Acronym: GUIDED-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Stony Brook University (Other); Indiana University (Other); Wayne State University (Other); VA Office of Research and Development (U.S. Federal Agency); University of Cincinnati (Other); Washington University School of Medicine (Other); Baylor College of Medicine (Other); MetroHealth Medical Center (Other); University of Mississippi Medical Center (Other); Emory University (Other); University of Iowa (Other); Thomas Jefferson University (Other); University of Texas (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Sean Collins, Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 150684
Record Dates: First submitted 2015-07-31; First posted 2015-08-10 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
Keywords: AHF; HF; ED; ER; Emergency Department; Emergency Room
MeSH Terms: conditions — Heart Failure; Emergencies | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): In keeping with the strategy-based pragmatic nature of the trial, the discharge procedures will largely be kept as they are in common practice. Investigators will standardize usual care for ED discharge to include HF medication reconciliation as well as encourage 7-day follow-up.
  Interventions: Behavioral: Standard of Care
- GUIDED-HF (Active Comparator): GWTG:HF has been successfully implemented across multiple inpatient populations and health systems over the last decade and has been shown to improve HF disparities.
  Interventions: Behavioral: GUIDED-HF

INTERVENTIONS:
Behavioral: GUIDED-HF — Participants in this arm will receive a tailored discharge plan via a transition nurse coordinator directed team (TNC Team).
  1. Disease education: Health literacy screen will identify barriers to understanding discharge and medication instructions.
  2. Lifestyle interventions: Includes receiving smoking cessation information and instructions to track daily weights.
  3. Guideline recommendations for medications and device referral: Includes determining the need for prescriptions for ACEIs, ARBs, beta blockers, aldosterone antagonists, anticoagulants and referral for pacemaker/defibrillator consideration.
  4. Outpatient follow-up appointment: TNC Team will provide a scheduled appointment within 7 days and will conduct a home visit within 48 hours of ED discharge.
  Arms: GUIDED-HF
Behavioral: Standard of Care — Those in the standard care arm will receive structured ED discharge assessment to include:
  1. discharge instructions;
  2. medication reconciliation
  3. encourage follow-up.
  Arms: Standard of Care

SUMMARY:
Approximately 20-30% of patients presenting with acute heart failure are discharged from the ED. Compared to patients discharged from the hospital, they more frequently return to the ED and hospital for further management. While inpatient discharges are often enrolled in transitions programs and have their care tailored to evidence-based recommendations, ED discharges do not. The investigators propose to evaluate current standard ED discharge to an ED-based intervention which will transition patients to outpatient follow-up on guideline-recommended therapy.

DETAILED DESCRIPTION:
Heart failure (HF) is common and growing healthcare concern. Heart failure affects nearly 6 million Americans. It results in over one million annual hospital discharges as the primary discharge diagnosis and an additional two million hospitalizations where HF contributes to the discharge diagnosis. Despite a relative reduction in the hospitalization rate of HF, the actual number of HF hospitalizations remains over one million annually. This figure is expected to significantly worsen with the aging United States population and the growing HF prevalence. Over 80% of patients who are hospitalized are initially seen in the emergency department (ED). However, not all those seen in the ED for HF are admitted; a sizeable proportion are discharged home without hospitalization. As disposition decisions for those who present to the hospital rest largely with ED providers, the ED will play an even bigger role in the management of HF patients and in avoiding unnecessary hospitalizations.

The ED is the gatekeeper for AHF evaluations. Nearly one million ED visits for acute heart failure (AHF) occur annually in the United States. Importantly, the ED is the safety net for AHF care and often sole provider of AHF care to vulnerable patients. To optimize care and reduce ED and hospital revisits, there has been significant emphasis on improving transitions at the time of hospital discharge for HF patients. Such efforts have been almost exclusively directed at hospitalized patients; individuals with AHF who are discharged from the ED miss the benefits of transitional care initiatives.

Ensuring optimal transitions of care for discharged ED AHF patients is a critical unmet need. Data show AHF patients discharged from the ED receive suboptimal guideline directed medical therapy (GDMT), suggesting interventions to improve AHF transitions are needed in the ED setting. This is particularly true for patients that are in resource limited settings, many of whom have vulnerable characteristics. By default the ED is often the sole or primary provider of HF care to this group of patients who are discharged from the ED.

The proposal, "Get with the Guidelines in ED Patients with Heart Failure (GUIDED-HF)", is designed to answer two fundamental questions about vulnerable patients with AHF discharged from the ED:

1. Does GWTG:HF implementation by a transition nurse coordinator directed team (TNC Team) reduce disparities in time to ED/clinic revisit or hospital admission or cardiovascular death over the 3-month period immediately following the index ED visit?
2. Does GWTG:HF implementation by a TNC Team reduce disparities in patient satisfaction, HF knowledge and QOL over the 3-month period immediately following the index ED visit?

Patients hospitalized for HF continue to have a high risk of adverse post-discharge outcomes. Although there has been a relative reduction in rehospitalization and mortality rates for AHF patients post-discharge after a significant recent effort by hospitals to avoid CMS financial penalties, the absolute risk remains very high. The one-month post discharge readmission risk is 20-25% and one-year post discharge mortality is 25-30%. These results are from institutions who have implemented significant in-hospital case management programs with a specific focus on transitions of care, including early post-discharge follow-up. ED patients discharged with AHF have more vulnerable characteristics, have a higher risk of readmission, and are not included in hospital programs targeted to help them. This proposal will study a significant unmet need, projected to get worse, and for which no evidence based data currently exist to guide management. Even a modest reduction in the risk for ED revisits or hospital admissions has the potential for significant clinical and patient centric benefits in patients with AHF discharged from the ED.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed by emergency physician to have AHF, who they plan to discharge or hold for brief ED-based observation (less than 23 hours of AHF care)
* Age ≥21 years old
* Prior history of HF

Exclusion Criteria:

* Unable to comply with protocol- due to psychiatric disease or distance from the hospital
* Systolic BP <100 mmHg
* Evidence of ACS based on ischemia on ECG or Troponin elevation
* Outpatient inotrope infusion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Composite Score Reflective of Clinical Status | 90 days from ED discharge
  Participants ranked sequentially. Ranking stratified in 1 of 3 tiers based on:
  Lowest tier: CV Death: Ranking based on time to death from original ED discharge date. Participant with the first death = lowest rank in the tier.
  Middle tier: ED Re-visit, Hospital Re-admission or Clinic for AHF with IV. For patients alive, ranking based on time to ED Re-visit, Hospital Re-admission or Clinic for AHF with IV from original ED discharge date, whichever occurs first. Participant with first adverse event = lowest rank in the tier.
  Highest tier: KCCQ Changes. For patients alive, ranking is based on changes in KCCQ from baseline. Participant with the largest decrease = lowest rank in the tier.
  The use of 3 tiers reflects the greater adverse impact of death, followed by adverse impact of Hospital Re-admission, ED Re-visit, clinic for AHF with IV on clinical status, and then health status as measured by KCCQ. The Clinical Events (Composite) updated on 11/19/19 per PCORI study team discussion.

SECONDARY OUTCOMES:
HF Related Quality of Life: Kansas City Cardiomyopathy Questionnaire (KCCQ) | Enrollment, 30 days and 90 days after ED discharge
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 12-item self-administered questionnaire developed to independently measure the patient's perception of their health status. Scores range from 0 to 100, with higher scores indicating lower symptom burden and better QOL. Scores were divided into ranges of 0 to 25 (severe), 26 to 50 (moderate), 51 to 75 (fair), and 76 to 100 (little-to-no disability).
Adherence to Refills and Medications Scale (ARMS 7) score | Enrollment, 30 days and 90 days after ED discharge
  The ARMS consists of 7 questions administered verbally by healthcare professionals to assess self-reported adherence to medication for participants. Scores range from 7 to 28 with lower scores indicating better adherence and higher scores indicating worse adherence.
Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety score | Enrollment, 30 days and 90 days after ED discharge
  The PROMIS Anxiety short form consists of 8 questions with five response options ranging in value from 1 to 5 to assess self-reported anxiety for participants. Scores range from 8 to 40. Higher scores indicate greater anxiety.
Patient Reported Outcomes Measurement Information System (PROMIS) Depression score | Enrollment, 30 days and 90 days after ED discharge
  The PROMIS Depression short form consists of 8 questions with five response options ranging in value from 1 to 5 to assess self-reported anxiety for participants. Scores range from 8 to 40. Higher scores indicate greater depression.
Time spent at clinic office visits | 30 days and 90 days after ED discharge
  Time spent at clinic office visits after ED discharge will be measured in minutes. Increased minutes indicate lower health status
Out-of-pocket costs for work missed | 30 days and 90 days after ED discharge
  Out-of-pocket costs for time missed at work after ED discharge will be measured in dollars. Increased dollars indicate lower health status
Dutch Heart Failure Knowledge score | Enrollment, 30 days and 90 days after ED discharge
  The Dutch Heart Failure Knowledge Scale is a 15-item, self-administered questionnaire that covers items concerning HF knowledge. Scores range from 0 to 15, where a score between 0 and 7 indicates a lack of awareness and a score between 8 and 15 indicates a complete knowledge of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Collins, MD, Principal Investigator — Vanderbilt University; Javed Butler, MD, Principal Investigator — Stony Brook University
Locations (15):
- United States (15):
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Stony Brook University, Stony Brook, New York
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - VA Tennessee Valley Health System, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Stubblefield WB, Jenkins CA, Liu D, Storrow AB, Spertus JA, Pang PS, Levy PD, Butler J, Chang AM, Char D, Diercks DB, Fermann GJ, Han JH, Hiestand BC, Hogan CJ, Khan Y, Lee S, Lindenfeld JM, McNaughton CD, Miller K, Peacock WF, Schrock JW, Self WH, Singer AJ, Sterling SA, Collins SP. Improvement in Kansas City Cardiomyopathy Questionnaire Scores After a Self-Care Intervention in Patients With Acute Heart Failure Discharged From the Emergency Department. Circ Cardiovasc Qual Outcomes. 2021 Oct;14(10):e007956. doi: 10.1161/CIRCOUTCOMES.121.007956. Epub 2021 Sep 24. PMID 34555929
- [Derived] Collins SP, Liu D, Jenkins CA, Storrow AB, Levy PD, Pang PS, Chang AM, Char D, Diercks DJ, Fermann GJ, Han JH, Hiestand B, Hogan C, Kampe CJ, Khan Y, Lee S, Lindenfeld J, Martindale J, McNaughton CD, Miller KF, Miller-Reilly C, Moser K, Peacock WF, Robichaux C, Rothman R, Schrock J, Self WH, Singer AJ, Sterling SA, Ward MJ, Walsh C, Butler J. Effect of a Self-care Intervention on 90-Day Outcomes in Patients With Acute Heart Failure Discharged From the Emergency Department: A Randomized Clinical Trial. JAMA Cardiol. 2021 Feb 1;6(2):200-208. doi: 10.1001/jamacardio.2020.5763. PMID 33206126
- [Derived] Fermann GJ, Levy PD, Pang P, Butler J, Ayaz SI, Char D, Dunn P, Jenkins CA, Kampe C, Khan Y, Kumar VA, Lindenfeld J, Liu D, Miller K, Peacock WF, Rizk S, Robichaux C, Rothman RL, Schrock J, Singer A, Sterling SA, Storrow AB, Walsh C, Wilburn J, Collins SP. Design and Rationale of a Randomized Trial of a Care Transition Strategy in Patients With Acute Heart Failure Discharged From the Emergency Department: GUIDED-HF (Get With the Guidelines in Emergency Department Patients With Heart Failure). Circ Heart Fail. 2017 Feb;10(2):e003581. doi: 10.1161/CIRCHEARTFAILURE.116.003581. PMID 28188268